

SAP Version: 1 CIP Version: 3

CIP Version Date: 27-APR-2022

### Statistical Analysis Plan (SAP)

#### FINS

| Clinical Investigation Title: | Lower Extremity Fixation In Neuropathic Patients Study (FINS) |
|---|---|
| Device Name: | HOFFMANN® LRF SYSTEM SALVATION™ EXTERNAL FIXATION SYSTEM SALVATION™ FUSION BOLTS AND BEAMS SALVATION™ 2 MIDFOOT NAIL SALVATION™ 3DI PLATING SYSTEM T2® ICF SYSTEM VALOR™ ANKLE FUSION NAIL SYSTEM |
| Clinical Investigation Plan<br>(CIP) Version: | 3 |
| Investigational Devices | HOFFMANN® LRF SYSTEM SALVATION™ EXTERNAL FIXATION SYSTEM SALVATION™ FUSION BOLTS AND BEAMS SALVATION™ 2 MIDFOOT NAIL SALVATION™ 3DI PLATING SYSTEM T2® ICF SYSTEM VALOR™ ANKLE FUSION NAIL SYSTEM |
| Indications | Detailed in the devices' Instructions for Use (IFU) and Surgical Technique Manual. |
| Clinical Investigation Design: | Prospective, observational, multi-site, multi-year post-market clinical follow-up study |
| Statistical Analysis Plan (SAP)<br>Version: | 1 |
| Date: | 14 – February- 2023 |
| Confidentiality Statement: | This Statistical Analysis Plan contains confidential information, and its' use is limited to investigational staff intending to conduct the clinical investigation, Institutional Review Boards (IRBs)/Ethics Committees (ECs) and any others charged with reviewing the clinical investigation. |




#### 1 Administrative Information

#### **Signatories and Approvers**

#### Prepared by:

| Role | Name, Title | Signature | Date |
|---|---|---|---|
| Author/<br>Statistician | Jovi Quiton<br>Senior Manager, Statistics | DocuSigned by: Myruth | 2/22/2023 |
| | | 74CDF10AA94943E | |

#### Reviewed by:

| Role | Name, Title | Signature | Date |
|---|---|---|---|
| Clinical Research Head (CRH) | <b>David Fitch</b><br>Director | David Fitch | 2/22/2023 |
| Clinical Investigation<br>Manager (CIM) | Monica Fleeman<br>Senior Clinical Study<br>Manager | E1459B1F4E7B4D1 Docusigned by: Monica Fleeman | 2/14/2023 |
| Clinical Operations Head (ClinOps) | <b>Rebecca Gibson</b> Director | 9D851D9B8FC415 DocuSigned by: Rebecce Gibson B69B71B0C1FA437 | 2/15/2023 |

SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

#### 2 Table of Contents

| 1 | Adn | ninistrative Information | 2 |
|---|------|--------------------------------------------------|----|
| 2 | Tab | le of Contents | 3 |
| 3 | List | of Abbreviations and Definitions | 5 |
| 4 | Intr | oduction | 7 |
| | 4.1 | Background and Rationale | 7 |
| | 4.2 | Clinical Investigation Purpose | 7 |
| 5 | Clin | ical investigation Objectives and Endpoints | 8 |
| | 5.1 | Primary Endpoints | 8 |
| | 5.2 | Secondary Endpoints | 8 |
| | 5.3 | Other Exploratory Endpoints | 8 |
| 6 | Clin | ical Investigation Methods | 8 |
| | 6.1 | General Clinical Investigation Design and Plan. | 8 |
| | 6.2 | Inclusion-Exclusion Criteria | 9 |
| | 6.3 | Withdrawal / Follow-up | 9 |
| | 6.4 | Methods to Minimize Bias and Confounding Factors | 9 |
| | 6.5 | Clinical Investigation Assessments | 9 |
| | 6.6 | Sample Size | 10 |
| 7 | Gen | eral Analysis Considerations | 10 |
| | 7.1 | Timing of Analyses | 10 |
| | 7.2 | Analysis Populations | 11 |
| | 7.3 | Covariates and Subgroups | 11 |
| | 7.4 | Multicenter Clinical investigations | 11 |
| | 7.5 | Missing Data | 11 |
| | 7.6 | Multiple Testing/Comparison | 11 |
| | 7.7 | Conventions | 11 |
| 8 | Sun | nmary of Clinical Investigation Data | 11 |
| | 8.1 | Subject Disposition | 11 |
| | 8.2 | Subject Accounting | 11 |
| | 8.3 | CIP Deviations | 11 |
| | 8.4 | Demographics and Disease pre-operative state | 12 |
| | 8.5 | Operative Variables | 12 |
| 9 | Sun | nmary of Effectiveness/Performance Data | 12 |

### *s*tryker

# Statistical Analysis Plan for FINS (US20-SAL-001)


| 9.1 | Primary Effectiveness/Performance Analysis | 13 |
|---|---|---|
| 9.2 | Analyses of Secondary Effectiveness Endpoints | 13 |
| 10 | Safety Analyses | 13 |
| 10.1 | Adverse Events | 13 |
| 10.2 | 2 Serious Adverse Events | 13 |
| 11 | Reporting Conventions | 14 |
| 12 | Summary of Changes to the CIP and/or SAP | 14 |
| 13 | Statistical Software | 14 |
| 14 | Listing of Tables, Listings, and Figures (TLF) | 14 |
| 14.1 | o de la companya de la companya de la companya de la companya de la companya de la companya de la companya de | |
| 14.2 | 2 Listing of Listings | 15 |
| 14.3 | B Listing of Figures | 15 |
| 15 | References and Related Documents. | 16 |
| 15.1 | All Table Shells | 17 |




#### 3 List of Abbreviations and Definitions

| Abbreviation | Explanation |
|---|---|
| AE(s) | Adverse Event(s) |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval |
| CIP | Clinical Investigation CIP |
| CRF | Case Report Form |
| EC | Ethics Committee |
| FU | Follow-Up |
| EDC | Electronic Data Capture |
| EQ-5D-5L | A standardized health-related quality of life instrument by the EuroQuol Group |
| FAAM-SANE | Foot and Ankle Ability Measure-Single Assessment Numeric Evaluation |
| FDA | Food and Drug Administration |
| ITT | Intend-to-Treat Population |
| IQR | Interquartile Range |
| KM | Kaplan-Meier |
| LOCF | Last Observation Carried Forward |
| MEDRA | Medical Dictionary for Drug Regulatory Affairs |
| N (or n) | Total Sample Size (or subgroup sample size) |
| PMA | Pre-Market Authorization |
| PMCF | Post-Market Clinical Follow-Up |
| PP | Per Protocol Population |
| PROM | Patient Reported Outcome Measures |
| QoL | Quality of Life |
| OR | Odds Ratio |
| RR | Relative Risk |
| SADE(s) | Serious Adverse Device Effect(s) |
| SAE(s) | Serious Adverse Event(s) |
| SAF | Safety Population |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| UADE(s) | Unanticipated Adverse Device Effect(s) |
| USADE(s) | Unanticipated Serious Adverse Device Effect(s) |




| Term | Definition |
|---|---|
| Adverse Event | Any untoward medical occurrence in patients/subjects, users or other persons. In the context of clinical investigation, for patients/subjects, |
| | this would include all untoward medical occurrences, whether or not |
| | related to the investigational device, that occurred in the course of the |
| | investigation. In the context of clinical experience, this would only |
| | include untoward medical occurrences that may be related to the |
| | medical device. |
| Clinical Performance | The ability of a medical device to achieve its intended clinical purpose as |
| | claimed by the manufacturer. |




#### 4 Introduction

#### 4.1 Background and Rationale

This statistical analysis plan is developed to provide the analytic framework and the production of statistical output of the FIN Study. This analysis plan is based on the FINS CIP version 3, dated 27 April 2022. The FIN Study was a prospective, multisite, multiyear, post-market follow-up clinical (PMCF) investigation that aimed to compare the pooled three-year amputation rate of the investigational devices in **Table 1** to a performance goal derived from a literature-based source. The study planned to enroll at least 200 subjects at 10 sites in the US, however, the Sponsor decided to discontinue the enrollment on 28 October 2022. Approximately 42 subjects were implanted with at least one investigational device when the study was discontinued. This statistical plan will guide the statistical analysis and presentation of these subjects that were enrolled and implanted with any of the devices under investigation.

Table 1. Study Device FDA 510K Clearance Information

| Device Name | Date of Clearance | 510K Number |
|----------------------------------------|-------------------|-------------|
| HOFFMANN® LRF SYSTEM | 01Feb2021 | K203568 |
| SALVATION™ EXTERNAL FIXATION<br>SYSTEM | 06Jun2018 | K180832 |
| SALVATION™ FUSION BOLTS AND BEAMS | 21Mar2014 | K140741 |
| SALVATION™ 2 MIDFOOT NAIL | 11Jul2018 | K180024 |
| SALVATION™ 3DI PLATING SYSTEM | 22May2014 | K140792 |
| SALVATION™ OSTEOPENIC SCREW | 14May2014 | K140408 |
| T2® ICF SYSTEM | 20Mar2020 | K193366 |
| VALOR™ ANKLE FUSION NAIL | 220ct2014 | K142602 |

#### 4.2 Clinical Investigation Purpose

The Sponsor identified a need to collect PMCF data to verify the safety and efficacy/performance of the HOFFMANN® LRF SYSTEM, SALVATION™ EXTERNAL FIXATION SYSTEM, SALVATION™ FUSION BOLTS AND BEAMS, SALVATION™ 2 MIDFOOT NAIL, SALVATION™ 3DI PLATING SYSTEM, T2® ICF SYSTEM, and VALOR™ ANKLE FUSION NAIL Systems. The study was initiated to demonstrate the safety and performance/efficacy of these systems using the data collected. The study planned to assess efficacy through the 3-year amputation rate. Safety was to be assessed through the incidence of device-related intra-operative and post-operative adverse events/incidents (AEs) by 5 years. The study planned to follow all subjects annually post-operatively for 5 years.




#### 5 Clinical investigation Objectives and Endpoints

The primary effectiveness hypothesis is that the 3-year amputation rate (including both above and below the knee) is less than the performance goal (PG).

#### 5.1 Primary Endpoints

The primary endpoint of the study was the overall performance of the devices (HOFFMANN® LRF SYSTEM, SALVATION™ EXTERNAL FIXATION SYSTEM, SALVATION™ FUSION BOLTS AND BEAMS, SALVATION™ 2 MIDFOOT NAIL, SALVATION™ 3DI PLATING SYSTEM, T2® ICF SYSTEM, and VALOR™ ANKLE FUSION NAIL Systems) measured as the 3-year amputation rate.

#### 5.2 Secondary Endpoints

The secondary performance endpoints were:

- Improvement in patient-reported function, and social interaction for quality of life via
  - EuroQuol five dimensions (EQ-5D-5L); and
  - o Foot and Ankle Ability Measure (FAAM).
- Performance or survival of the device measured as the 5-year Amputation Rate

The secondary safety endpoints were:

- incidence and rate of AEs through 5 years;
- physical and radiographic assessment of the implant status; and
- rate of surgical Intervention

#### 5.3 Other Exploratory Endpoints

None

#### 6 Clinical Investigation Methods

This investigation was a prospective, multicenter PMCF study. The clinical investigation was designed to follow the surgeon's standard of care for the treatment of deformity in the neuropathic patient over 5 years.

#### 6.1 General Clinical Investigation Design and Plan

This study was designed to clinically assess over time the effectiveness and safety of the devices under investigation. There was no randomization of subjects employed. The study did not employ any methods (e.g., randomization, blinding, or stratification) for assigning subjects. Consecutive subjects at each site that met all the eligibility criteria were invited to enroll in the study. The study planned to collect data from subjects before implant surgery, during the procedure, 6 months post-operative and annually thereafter for five years. Demographic factors, Medical History, and disease state were collected at baseline. The patient-reported outcomes, EQ-5D-5L and FAAM were collected at baseline, at 6 months post-operative and at scheduled annual post-surgery visits to evaluate improvement in pain, function, social interaction, and quality of life. Safety of the implants in terms of complications and adverse events that occurred during the study was collected.




#### 6.2 Inclusion-Exclusion Criteria

Subjects that met the following inclusion criteria were invited to be enrolled in the study.

- a. Subject was a male or non-pregnant female age 18 years or older at the time of surgery;
- b. Subject was willing and able to give written informed consent and comply with the requirements of the Clinical Investigation Plan (CIP); and
- c. Subject had neuropathy and intended to be treated for deformity with the one or a combination of the below Systems in accordance with the legally cleared/approved IFU and Surgical Technique Manual.
  - HOFFMANN® LRF SYSTEM
  - SALVATION™ EXTERNAL FIXATION SYSTEM
  - SALVATION™ FUSION BOLTS AND BEAMS
  - SALVATION™ 2 MIDFOOT NAIL
  - SALVATION™ 3DI PLATING SYSTEM
  - o T2® ICF SYSTEM
  - VALOR™ ANKLE FUSIO NAIL SYSTEM

#### Subjects that were

- a. determined, by the investigator, to be an inappropriate candidate for the procedure indicated; or
- b. unable to consent to participate (written, informed consent); or
- c. unable to attend/complete the requested follow-up visits

were excluded from the study

#### 6.3 Withdrawal / Follow-up

The study allowed subjects to withdraw from the clinical investigation for any of the following reasons:

- a. Voluntary withdrawal by the subject;
- b. Subject was Lost to Follow-Up (LTFU);
- c. Amputation below the knee or above the knee;
- d. Adverse event that prohibited the subject from continued participation;
- e. Subject non-compliance to study protocol; and
- f. Other reason(s) that may have exposed the subject to unacceptable risk.

#### **6.4** Methods to Minimize Bias and Confounding Factors

The study design did not employ a method for assigning subjects. A consecutive series of subjects at each site meeting all the eligibility criteria were enrolled in the study.

#### **6.5 Clinical Investigation Assessments**

The study collected subject data at baseline, surgery, 6 months, 1 year, and at 2-5 years post-surgery follow-up visits. The follow-up evaluations included the patient-reported outcome measures: EQ-5D-5L and FAAM, adverse events, and occurrence of surgical intervention. Refer to **Table 2** below for the visit windows and the list of assessments performed at each visit as indicated in the CIP. There will be no windowing of days elapsing from surgery to a visit date and the determination of post-operative visit will be based on the visit completed indicated in the study form.




Table 2. Schedule of Events

| Assessment | Pre-<br>Operative | Operative/<br>Discharge | 6 months a, b<br>(+/-3<br>months) | 1 Year <sup>a,b</sup><br>(+/-6 months) | 2-5 years <sup>a, b</sup><br>(+/-6 months) | Study<br>Close |
|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | |
| Inclusion/Exclusion | X | | | | | |
| Demographics &<br>Medical History | X | | | | | |
| Disease State Pre-Op | X | | | | | |
| EQ-5D-5L | X | | X | X | X | |
| FAAM | X | | X | X | X | |
| Surgical Procedure | | X | | | | |
| Investigator Assessment | | | X | X | X | |
| Adverse Event<br>Assessment | | X | X | X | X | |
| Staged Operative Information <sup>d</sup> | | | | | | |
| Surgical Intervention d | | | | | | |
| Subject Disposition c | | | | | | X |

- a. Follow-up visit schedule to reflect Institutions' Standard of Care practices.
- b. If the subject missed a visit and is outside of visit window, every effort should be made to collect data instead of noting visit as missed.
- c. Subject Disposition assessment will occur at any time point for subject withdrawal prior to the completion of the clinical investigation.
- d. These are not scheduled time point events but will be observed throughout the study participation

#### 6.6 Sample Size

The study required a sample size of 141 patients to provide at least 80% statistical power to reject the hypothesis that the 3-year amputation rate is less than the PG with a significance  $\alpha$ =0.05. However, this sample size requirement was not met at to study discontinuation.

#### 7 General Analysis Considerations

Data will be summarized for each of the devices listed in **Table 1**. Because the study was prematurely terminated, all analysis will be descriptive only. All analyses will be done to summarize all available data. No statistical hypothesis testing will be implemented.

#### 7.1 Timing of Analyses

Statistical summaries will be implemented for the final data, that is, all data collected in the study.




#### 7.2 Analysis Populations

All subjects who received any clinical investigation treatment/device upon study termination are included in the ITT and safety population.

#### 7.3 Covariates and Subgroups

No subgroup analysis will be conducted.

#### 7.4 Multicenter Clinical investigations

Except for the study site distribution of subjects, no center specific analysis will be conducted.

#### 7.5 Missing Data

No imputation of missing data will be conducted.

#### 7.6 Multiple Testing/Comparison

No test of hypothesis will be conducted.

#### 7.7 Conventions

In the case of collection of variables with non-SI units (e.g., pounds instead of kilograms), conversion of such data into SI units (and vice versa) will be ensured. The data for both SI and non-SI units will be reported in the final listing of data. Differences between score results will be calculated.

#### 8 Summary of Clinical Investigation Data

The statistical analysis will be implemented to summarize the data collected upon study termination. All data will be summarized by visit and by device, whenever possible. Categorical and ordinal data will be displayed as frequency and percent. Continuous data will be summarized with the following summary statistics (number of observations, mean, median, standard deviation, inter-quartile range, minimum, and maximum).

#### 8.1 Subject Disposition

Distribution of subjects by investigational device and overall will be presented. Also, the site distribution of subjects by, visit completion and the reason for study non-completion will be presented.

#### 8.2 Subject Accounting

The subject accounting will present the frequency of subjects that are expected for follow-up, the rate of actual follow-up and the assessment of visit compliance.

#### 8.3 CIP Deviations

The extent of protocol deviations that occurred in the study will be presented. CIP deviations that could impact the analysis will not be assessed.



SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

#### 8.4 Demographics and Disease pre-operative state

The demographic factors: gender (M/F), age (years), smoking status, body mass index (BMI), race, diabetes status, and disease state. Pre-operative disease state variables included: Brodsky/Trepman Classification, Pre-operative state (walking or with aids), pain level, presence of a chronic ulcer, infection, insulin use, type peripheral neuropathy, revascularization history, peripheral artery disease retinopathy, and chronic kidney disease.

#### 8.5 Operative Variables

The following surgical information will be summarized: indication for implant use, operative side (left or right), previous surgery to index procedure, biologics use, and intraoperative complications.

#### 9 Summary of Effectiveness/Performance Data

#### EuroQol (EQ-5D-5L)

A generic health survey can be used to compare improvement across different interventions and measure changes in health-related quality of life over time. The EQ-5D-5L comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and 100 on VAS indicates the best health, whereas 0 on the VAS indicates the worst health. Patient health profiles with concerning mobility, self-care, activities, pain/discomfort and anxiety/depression will be presented as frequency and rates. In addition, the summaries for improvement from baseline in VAS health score will be presented. Also, summaries for the converted EQ-5D-5L index value will be presented. At each post-surgery follow-up visit, descriptive statistics and confidence interval estimates of the mean will be constructed for the change in scores.

#### **FAAM**

The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument to assess physical function for individuals with foot and ankle-related impairments. The FAAM consists of 29-item questions divided into two subscales: 21-item activities of daily living (ADL) subscale, an 8-item sports subscale. Each item is scored on a 5-point Likert scale (4 to 0) from 'no difficulty at all' to 'unable to do'. Responses of "not applicable" are not counted. The scores of the sub-scale items will be added together to get the subscale total score. The ADL subscale total score ranges from 0 to 84, and 0 to 32 for the sports subscale. The patient score for the ADL and sports subscale will be transformed into percentage scores by considering the highest possible score for non-missing items. A higher score indicates a higher level of function for each subscale, with 100% representing no dysfunction (Martin et al., 2009).

#### Surgeon Assessment and radiographic outcome

The attending surgeon assessed the outcome of the implant one year after surgery and at the final visit. The following factors were assessed by the surgeon:

- Insulin use
- Ulcer healing and presence of new ulcers
- Presence of new deep infection
- Ankle alignment status
- Current mobility status (walking, use of mobility aids)



SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

on version bace. 27 in it 2022

In addition, radiographic assessment of deformity correction was collected. The surgeon assessment of angle deformity correction based on radiograph will be summarized for the following:

- Meary's angle deformity: Lateral & AP;
- Talonavicular angle; and
- Cuboid height (mm)

#### 9.1 Primary Effectiveness/Performance Analysis

None of the subjects reached their three-year post-surgery follow-up. Thus, the three-year amputation rate, which is the primary endpoint will not be analyzed. Instead, the frequency of amputations at each post-surgery visit will be presented. The status of the subject at the latest follow-up, coded as either walking, use of mobility aids, bedridden or having amputation will be summarized instead.

#### 9.2 Analyses of Secondary Effectiveness Endpoints

EQ-5D-5L and FAAM scores will be summarized at each visit. In addition, score improvement at each post-operative visit will also be summarized by the change from baseline score in EQ-5D-5L and FAAM total and their component scores. Also, the post-operative physical and radiographic assessment of the surgical foot and the implant by the investigator will be summarized.

#### 10 Safety Analyses

The safety data will be summarized by the frequency and percentage of AE incidence. Each AE was also assessed according to the relationship to the clinical investigation device and severity.

#### 10.1 Adverse Events

The safety of each device will be summarized in the final report. The overall summary of adverse events will be presented for each device. Total events, patient counts and percentages of adverse events for each device will be summarized for the following factors:

- i.) Procedure-Related Adverse Event / Incident.
- ii.) Device-Related Adverse Event / Incident
- iii.) Device Failure
- iv.) Serious Adverse Event (SAE)
- v.) Hospitalization SAE Outcome
- vi.) Treatment Required for the AE

#### 10.2 Serious Adverse Events

A separate summary table (or listing) of complications that met the serious adverse events (SAE) classification will be presented. Also, this section presents the narratives of each SAE that occurred in the clinical investigation. A serious adverse event (SAE) as defined from ISO 14155:2020(E) Clinical Investigations of Medical Devices for Human Subjects – Good clinical practice, is any adverse event that:

a. Led to death,

b. Led to a serious deterioration in the health of the subject, that either resulted in




- A life-threatening illness or injury, or
- A permanent impairment of a body structure or a body function, or
- In-patient or prolonged hospitalization, or
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.

c. Led to fetal distress, fetal death or congenital abnormality or birth defect.

The narrative for each SAE will be presented to describe the following:

- Nature and intensity of the event,
- Clinical course leading up to the event,
- Indication of timing relevant to test investigational device/product administration,
- Relevant laboratory measurements;
- Whether the treatment was stopped, and countermeasures (and timing);
- Post-mortem findings;
- Investigator's opinion on causality and sponsor's opinion on causality, if appropriate.

In addition, the following information will be included (if available) in the SAE narrative:

- Patient identifier:
- Age and sex of patient; general clinical condition of the patient, if appropriate;
- Disease being treated (this is not required if it is the same for all patients) with duration (of the current episode) of illness;

#### 11 Reporting Conventions

All statistical output will have the following standard elements:

| Stryker Corporation US-20-SAL-001-FINS | Title of Display<br>Clinical investigation Population<br><body display="" of=""></body> | Page of |
|---|---|---|
| Data Version: <date9> Execution date: <date9> Listing Reference: <listing #=""></listing></date9></date9> | | <pre><pre><pre><pre>ogram name&gt;</pre></pre></pre></pre> |

#### 12 Summary of Changes to the CIP and/or SAP

No changes to the planned statistical analysis as indicated in the CIP.

#### 13 Statistical Software

All statistical analyses will be performed using SAS version 14.1 or higher.

#### 14 Listing of Tables, Listings, and Figures (TLF)

The listings of TLF are provided below with the link to the corresponding Table templates in Appendix 1.




#### **14.1 Listing of Tables**

| Table # | Table Title |
|------------------|------------------------------------|
| <u>Table 1.1</u> | Subject Disposition |
| <u>Table 1.2</u> | Subject Eligibility |
| <u>Table 1.3</u> | Subject Accounting |
| <u>Table 1.4</u> | CIP Deviations |
| <u>Table 1.5</u> | Demographic and Baseline Variables |
| <u>Table 1.6</u> | Medical History at Screening |
| <u>Table 1.7</u> | Pre-operative Disease State |
| Table 2.1 | Operative Information |
| <u>Table 3.1</u> | EQ-5D Score |
| <u>Table 3.2</u> | FAAM Score |
| <u>Table 3.3</u> | Surgeon Assessment |
| <u>Table 3.4</u> | Surgeon Radiographic Assessment |
| Table 4.1 | Summary of All Adverse Events |
| Table 4.2 | Device-related Adverse Events |
| Table 4.3 | Serious Adverse Events |

#### 14.2 Listing of Listings

| Listing # | Listing Title |
|------------|------------------------------------|
| Listing 1 | Subject Disposition |
| Listing 2 | CIP Deviations |
| Listing 3 | Subject Eligibility |
| Listing 4 | Demographic and Baseline Variables |
| Listing 5 | Medical History |
| Listing 6 | Pre-operative Disease State |
| Listing 7 | Operative Information |
| Listing 8 | Surgeon Physical Assessment |
| Listing 9 | Radiographic Assessment |
| Listing 10 | EQ-5D |
| Listing 11 | FAAM |
| Listing 12 | Adverse Events |

#### **14.3** Listing of Figures

No figures will be presented.




#### 15 References and Related Documents

Domsic RT, Saltzman CL. Ankle osteoarthritis scale. Foot Ankle Int. 1998; 19:466-471 EQ5D-5L Questionnaire; EQ-5D<sup>m</sup> is a trade mark of the EuroQol Research Foundation.

Maher, A, Kilmartin, T. An analysis of Euroqol EQ5D and Manchester Oxford Foot Questionnaire. *Journal of Foot and Ankle Research* 2012; 5; 7

Martin RL, Hutt DM, Wukich DK. Validity of the Foot and Ankle Ability Measure (FAAM) in Diabetes Mellitus. Foot Ankle Int. 2009 Apr;30(4):297-302

Lower Extremity Fixation In Neuropathic Patients Study (FINS) Clinical Investigation Plan Protocol. Version 2. 11-MAR-2022

Lower Extremity Fixation In Neuropathic Patients Study (FINS) Clinical Investigation Plan. Version 3 27-APR-2022



SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

#### 15.1 All Table Shells

**Table 1.1 Subject Disposition - ITT** 

| Device | Pre-Op | Final F-up<br>(Op- 1yr) | Post-Op<br>(1 yr.) |
|---|---|---|---|
| SALVATION™ 3Di Plating | I | (OP 191) | (1 )11) |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |
| SALVATION™ External Fixation | | | |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |
| SALVATION™ Fusion Bolts and Beam | S | | |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |
| SALVATION™ MIDFOOT NAIL | | | |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |




| Device | Pre-Op | Final F-up<br>(Op- 1yr) | Post-Op<br>(1 yr.) |
|---|---|---|---|
| VALOR™ Nail | | | |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |
| HOFFMANN® LRF SYSTEM | | | |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |
| T2® ICF SYSTEM | | | |
| Total | | | |
| Available Data | | | |
| Reason for Discontinuation | | | |
| Subject lost to follow-up | | | |
| Subject withdrew consent | | | |
| Adverse Event | | | |
| Other | | | |




#### **Table 1.2 Subject Eligibility**

| | Inclusion<br>Questions | | | Exclusion<br>Questions | | | Eligible |
|---|---|---|---|---|---|---|---|
| | 1 | 2 | 3 | 1 | 2 | 3 | |
| All Subjects | | | | | | | |
| By Device | | | | | | | |
| SALVATION™ 3Di Plating | | | | | | | |
| SALVATION™ Fusion Bolts and | | | | | | | |
| Beams | | | | | | | |
| SALVATION™ External Fixation | | | | | | | |
| SALVATION™ MIDFOOT NAIL | | | | | | | |
| <b>VALOR™ Nail</b> | | | | | | | |
| Total | | | | | | | |

Note:

**Inclusion 1** - Subject is a male or non-pregnant female age 18 years or older at the time

**Inclusion 2** - Subject is willing and able to give written informed consent and comply with the requirements of this Clinical Investigation Plan (CIP); and

**Inclusion 3** - Subject has or is intended to be treated for neuropathy with the one or a combination of the below Systems in accordance with the legally cleared/approved IFU and Surgical Technique Manual.

- o HOFFMANN® LRF SYSTEM
- o SALVATION™ EXTERNAL FIXATION SYSTEM
- o SALVATION™ FUSION BOLTS AND BEAMS
- o SALVATION™ 2 MIDFOOT NAIL
- o SALVATION™ 3DI PLATING SYSTEM
- o T2® ICF SYSTEM
- o VALOR™ ANKLE FUSIO NAIL SYSTEM

**Exclusion 1** – Subjects determined, by the investigator, to be an inappropriate candidate for the procedure indicated;

**Exclusion 2** - Unable to consent to participate (written, informed consent);

Exclusion 3 - Unable to attend/complete the requested follow-up visits




Table 1.3 Subject Accounting and Follow-up Compliance - ITT

| ınting and Follow-up Compliance - ITT | | 1 Year | Final Visit |
|---------------------------------------|-------------|--------|-------------|
| Device | Pre-op<br>N | N | N N |
| SALVATION™ 3Di Plating System | 14 | 14 | - 11 |
| Theoretical | | | |
| Deaths (cumulative) | | | |
| Failures (cumulative) | | | |
| Withdrawn (cumulative) | | | |
| Expected | | | |
| Actual <sup>1</sup> | | | |
| % Follow-up <sup>1</sup> | | | |
| EQ-5D Score | | | |
| FAAM Score | | | |
| SALVATION™ External Fixation | | | |
| Theoretical | | | |
| Deaths (cumulative) | | | |
| Failures (cumulative) | | | |
| Withdrawn (cumulative) | | | |
| Expected | | | |
| Actual <sup>1</sup> | | | |
| % Follow-up <sup>1</sup> | | | |
| EQ-5D Score | | | |
| FAAM Score | | | |
| SALVATION™ Fusion Bolts and Beams | | | |
| Theoretical | | | |
| Deaths (cumulative) | | | |
| Failures (cumulative) | | | |
| Withdrawn (cumulative) | | | |
| Expected | | | |
| Actual <sup>1</sup> | | | |
| % Follow-up <sup>1</sup> | | | |
| EQ-5D Score | | | |
| FAAM Score<br>SALVATION™ MIDFOOT NAIL | | | |
| Theoretical | | | |
| Deaths (cumulative) | | | |
| Failures (cumulative) | | | |
| Withdrawn (cumulative) | | | |
| Expected | | | |
| Actual <sup>1</sup> | | | |
| % Follow-up <sup>1</sup> | | | |
| EQ-5D Score | | | |
| FAAM Score | | | |
| VALOR™ Nail | | | |
| Theoretical | | | |
| Deaths (cumulative) | | | |
| Failures (cumulative) | | | |




| Withdrawn (cumulative) |
|----------------------------------------------------|
| Expected |
| Actual <sup>1</sup> |
| % Follow-up <sup>1</sup> |
| EQ-5D Score |
| FAAM Score |
| <sup>1</sup> Any data point available at follow-up |



SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

**Table 1.4 CIP Deviations** 

| | Dev 1 | Dev 2 | Dev 3 | Dev 4 | <b>Total Deviations</b> |
|---|---|---|---|---|---|
| All Subjects (N=114) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| SALVATION™ 3Di Plating | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| System | | | | | |
| SALVATION™ External | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| Fixation | | | | | |
| SALVATION™ Fusion Bolts | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| and Beams | | | | | |
| SALVATION™ MIDFOOT NAIL | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |
| VALOR™ Nail | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | XX |




**Table 1.5 Demographic and Baseline Variables** 

| Factors | Freq(%) |
|----------------------------------|------------|
| Gender | |
| Male | xx(xx.xx%) |
| Female | xx(xx.xx%) |
| Race | |
| African-American/Black | xx(xx.xx%) |
| Asian | xx(xx.xx%) |
| Hispanic/Latino | xx(xx.xx%) |
| Native American/Alaskan | xx(xx.xx%) |
| Native Hawaiian/Pacific Islander | xx(xx.xx%) |
| White | xx(xx.xx%) |
| Other | xx(xx.xx%) |
| Smoking Status | |
| Never | xx(xx.xx%) |
| Previous | xx(xx.xx%) |
| Current, <= 1 Pack/day | xx(xx.xx%) |
| Current, > 1 pack/day | xx(xx.xx%) |

| Factors | n | mean | std | min | max | median (IQR) | 95% CI |
|---|---|---|---|---|---|---|---|
| Age at Rx (years) | XX | XX.XX | XX.XX | XX.X | XX.X | xx.x(xx.x,xx.x) | (xx.x,xx.x) |
| Height (cm) | XX | XX.XX | XX.XX | XX.X | XX.X | xx.x(xx.x,xx.x) | (xx.x,xx.x) |
| Weight (kg) | XX | XX.XX | XX.XX | XX.X | XX.X | xx.x(xx.x,xx.x) | (xx.x,xx.x) |
| BMI (kg/m) | XX | XX.XX | XX.XX | XX.X | XX.X | xx.x(xx.x,xx.x) | (xx.x,xx.x) |




**Table 1.6 Medical History at Screening** 

| | All Subjects |
|-----------------------------------|--------------|
| | N=xx |
| Any Concomitant Health Conditions | |
| No | xx(xx.xx%) |
| Yes | xx(xx.xx%) |
| Autoimmune | xx(xx.xx%) |
| Cardiovascular | xx(xx.xx%) |
| Respiratory | xx(xx.xx%) |
| Gastrointestinal | xx(xx.xx%) |
| Hematological | xx(xx.xx%) |
| Psychological | xx(xx.xx%) |
| Musculoskeletal | xx(xx.xx%) |
| Neurological | xx(xx.xx%) |
| Endocrine | xx(xx.xx%) |
| Skin/Subcutaneous Tissue | xx(xx.xx%) |
| Peripheral Vascular Disease | xx(xx.xx%) |
| Diabetes | |
| Type I | xx(xx.xx%) |
| Type II | xx(xx.xx%) |
| Other Health Conditions | |
| No | xx(xx.xx%) |
| Yes | xx(xx.xx%) |



SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

**Table 1.7 Pre-operative Disease State** 

| | SALVATION™ | SALVATION™ | SALVATION™ | SALVATION™ | VALOR™ Nail |
|---|---|---|---|---|---|
| | 3Di Plating | External | Fusion Bolts and | MIDFOOT NAIL | (N=xx) |
| | (N=xx) | Fixation | Beams | (N=xx) | |
| | | (N=xx) | (N=xx) | | |
| Brodsky/Trepman Classification | | | | | |
| Type 1: Midfoot | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Type 2: Hindfoot | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Type 3a: Ankle | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Type 3b: Calcis tubercle | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Type 4: Combination | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Type 5: Forefoot | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Pre-operative state | | | | | |
| Walking with | | | | | |
| Custom shoes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Bracing | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| CROW boots | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Other | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Aids | | | | | |
| None | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Cane | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Walker | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Knee scooter | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Level of Pain | | | | | |
| mean±sd | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x | xx.x±xx.x |
| Ulcer | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Chronic Ulcer | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Deep Infection | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Insulin use | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Peripheral neuropathy, type | | | | | |
| Congenital | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Diabetes Mellitus | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Idiopathic/Unknown | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Post-Traumatic | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Peripheral artery disease | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| History of revascularization | | | | | |




| | SALVATION™ | SALVATION™ | SALVATION™ | VALOR™ Nail |
|---|---|---|---|---|
| 3Di Plating | External | Fusion Bolts and | MIDFOOT NAIL | (N=xx) |
| (N=xx) | Fixation | Beams | (N=xx) | |
| | (N=xx) | (N=xx) | | |
| xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| | (N=xx) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) | 3Di Plating (N=xx) External Fixation (N=xx) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) | 3Di Plating (N=xx) External Fixation (N=xx) Fusion Bolts and Beams (N=xx) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) | 3Di Plating (N=xx) External Fixation (N=xx) Fusion Bolts and (N=xx) MIDFOOT NAIL (N=xx) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) xx(xx.xx%) |




**Table 2.1 Operative Information** 

| | ORTHOLOC™ | SALVATION™ | SALVATION™ | SALVATION™ | <b>VALOR™ Nail</b> |
|---|---|---|---|---|---|
| | 3Di | External | <b>Fusion Bolts</b> | MIDFOOT NAIL | (N=xx) |
| | Midfoot/Flatfo | Fixation | and Beams | (N=xx) | |
| | ot | (N=xx) | (N=xx) | | |
| Indications for Use | | | | | |
| Post traumatic | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Arthritis | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Fracture | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Fusion | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Reconstruction/Correction | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Revision procedure | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Instability | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Skeletal defect | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Previous Surgery to Index procedure | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Operative Side | | | | | |
| Left | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Right | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Wright Biologics use | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Intra-operative complication | | | | | |
| No | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |
| Yes | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) | xx(xx.xx%) |



SAP Version: 1 CIP Version: 3 CIP Version Date: 27-APR-2022

Table 3.1 EQ-5D Score

| | | 1 | Baseline | | | Ē | Final Visit | | | 1 Y | 1 Yr. Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | u | Mean ± SD | min,max | 65% CI | u | Mean ± SD | min,max | 13 %56 | u | Mean ± SD | min,max | 95% CI |
| SALVATION™ Fusion Bolts and Beams | sion l | <b>Bolts and Bear</b> | ms | | | | | | | | | |
| EQ-VAS Score | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | xx.x, xx.x | XX.X, XX |
| EQ-5D Index | XX | $XX.X \pm XX.X$ | XXXX, XXXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XXX, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| EQ-VAS Score | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| EQ-5D Index | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| SALVATION™ MIDFOOT NAIL | DF0( | )T NAIL | | | | | | | | | | |
| EQ-VAS Score | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XXX, XXX | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX |
| EQ-5D Index | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| <b>EQ-VAS Score</b> | | | | | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XXX, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| EQ-5D Index | | | | | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XXX, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| SALVATION™ 3Di Plating System | i Plat | ting System | | | | | | | | | | |
| EQ-VAS Score | XX | $XX.X \pm XX.X$ | XXXX, XXXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XXX, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| EQ-5D Index | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| EQ-VAS Score | | | | | XX | XX.X ± XX.X | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX |
| EQ-5D Index | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| VALOR™ Nail | | | | | | | | | | | | |
| EQ-VAS Score | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| EQ-5D Index | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| EQ-VAS Score | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| EQ-5D Index | | | | | XX | $XXX \pm XXX$ | XX.X, XX.X | XXX, XXX | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX |
| SALVATION™ External Fixation | terna | Il Fixation | | | | | | | | | | |
| EQ-VAS Score | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX |
| EQ-5D Index | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| <b>EQ-VAS Score</b> | | | | | XX | XXX ± XXX | XX.X, XX.X | XX.X, XX.X | XX | XX.X ± XX.X | XX.X, XX.X | XX.X, XX |
| EQ-5D Index | | | | | XX | XX.X ± XX.X | XX.X, XX.X | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX |



Table 3.2 FAAM Score

| | | | Baseline | | | | Final Visit | | | 1 Y | 1 Vr. Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | u | Mean ± SD | min,max | 13 % 26 | u | Mean ± SD | min,max | 13 %56 | u | Mean ± SD | min,max | 95% CI |
| SALVATION™ Fusion Bolts and Beams | sion | <b>Bolts and Bea</b> | ms | | | | | | | | | |
| FAAM SANE | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $X.XX \pm X.XX$ | XXX, XXX | XX.X, XX |
| Sports Subscale | XX | $XX.X \pm XX.X$ | XXX, XXXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $X:XX \pm X:XX$ | XXX, XXX | XX.X, XX |
| ADL Subscale | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $X.XX \pm X.XX$ | XXX, XXX | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| FAAM SANE | | | | | XX | $X.XX \pm X.XX$ | XX.X, XX.X | XX.X, XX.X | XX | $X:XX \pm X:XX$ | XXX, XXX | XX.X, XX |
| Sports Subscale | | | | | XX | $X.XX \pm X.XX$ | XX.X, XX.X | XX.X, XX.X | XX | $X \cdot X \times $ | XXX, XXX | XX.X, XX |
| ADL Subscale | | | | | XX | $X.XX \pm X.XX$ | XX.X, XX.X | XX.X, XX.X | XX | $X'XX \mp X'XX$ | XXX, XXX | XX.X, XX |
| SALVATION™ MIDFOOT NAII | DFO | OT NAIL | | | | | | | | | | |
| FAAM SANE | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | Xx | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX |
| Sports Subscale | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | xx.x, xx.x | XX.X, XX |
| ADL Subscale | XX | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $X.XX \pm X.XX$ | XXX, XXX | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| FAAM SANE | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | xx.x, xx.x | XX.X, XX |
| Sports Subscale | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | xx.x, xx.x | XX.X, XX |
| ADL Subscale | | | | | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | X | $XX.X \pm XX.X$ | XXX, XXX | XX.X, XX |
| SALVATION™ 3Di Plating System | i Pla | ting System | | | | | | | | | | |
| FAAM SANE | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $XXX \pm XXX$ | XX.X, XX.X | XX.X, XX.X | XX | $XXX \pm XXX$ | XX.X, XX.X | XX.X, XX |
| Sports Subscale | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $XXX \pm XXX$ | XXX, XXX | XX.X, XX |
| ADL Subscale | XX | $XX.X \pm XX.X$ | XXX, XXXX | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $X:XX \pm X:XX$ | XXX, XXX | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| FAAM SANE | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | xxx, xxx | XX.X, XX |
| Sports Subscale | | | | | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| ADL Subscale | | | | | XX | $X.XX \pm X.XX$ | XX.X, XX.X | XX.X, XX.X | XX | $X:XX \pm X:XX$ | XXX, XXX | XX.X, XX |
| VALOR™ Nail | | | | | | | | | | | | |
| FAAM SANE | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $XXX \pm XXX$ | XX.X, XX.X | XX.X, XX.X | XX | $X:XX \pm X:XX$ | XXX, XXX | XX.X, XX |
| Sports Subscale | X | $xx.x \pm xx.x$ | XXX, XXX | XXX, XXX | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX |
| ADL Subscale | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $xx.x \pm xx.x$ | XXX, XXX | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| FAAM SANE | | | | | XX | $xx.x \pm xx.x$ | XXX, XX.X | XX.X, XX.X | XX | XX.X ± XX.X | XXX, XX.X | XX.X, XX |

# stryker

# Statistical Analysis Plan for FINS (US20-SAL-001)

| | | | Baseline | | | F | Final Visit | | | 1 Y | 1 Yr. Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | u | <b>Mean ± SD</b> | min,max | ID %56 | u | Mean ± SD | min,max | 95% CI | u | Mean ± SD | min,max | 95% CI |
| Sports Subscale | | | | | XX | $X.X. \pm X.X.$ | XX.X, XX.X | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| ADL Subscale | | | | | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | xx | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| SALVATION™ External Fixation | terna | l Fixation | | | | | | | | | | |
| FAAM SANE | XX | $XX.X \pm XX.X$ | XXXX, XXXX | XXXX, XX.X | XX | $XXX \pm XXX$ | XX.X, XX.X | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| Sports Subscale | XX | $XXX \pm XXX$ | XXX, XXXX | xxx, xxx | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX.X | XX | $XX.X \pm XX.X$ | xx.x, xx.x | XX.X, XX |
| ADL Subscale | XX | $XXX \pm XXX$ | XXX, XXX | XXX, XXX | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | xx | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| Change from Baseline | eline | | | | | | | | | | | |
| FAAM SANE | | | | | XX | XXX ± XXX | XX.X, XX.X | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| Sports Subscale | | | | | XX | XXX ± XXX | XX.X, XX.X | XXX, XX.X | XX | $xx.x \pm xx.x$ | XX.X, XX.X | XX.X, XX |
| ADL Subscale | | | | | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX.X | XX | $XX.X \pm XX.X$ | XX.X, XX.X | XX.X, XX |
| SANE -Single Assessment Numeric Evaluation. | ssmei | ıt Numeric Eva | luation. | | | | | | | | | |




**Table 3.3 Surgeon Assessment** 

| Device | Factors | 1 Yea | r Visit | Fina | l Visit |
|---|---|---|---|---|---|
| | | N | % | N | % |
| SALVATION™ Fusion Bolts<br>and Beams | Insulin Use | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ulcers | New | Ulcer | Ulcer | Healing |
| | Yes | XX | xx.x% | XX | xx.x% |
| | No | XX | xx.x% | xx | xx.x% |
| | Chronic Ulcer | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | New Deep Infection | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ankle Alignment | | | | |
| | Acceptable | | | XX | xx.x% |
| | Unacceptable | | | XX | xx.x% |
| | Not applicable | | | XX | xx.x% |
| | <b>Current Status</b> | | | | |
| | Walking | XX | xx.x% | XX | xx.x% |
| | Mobility with aids | XX | xx.x% | XX | xx.x% |
| | Wheelchair | XX | xx.x% | XX | xx.x% |
| | Bed ridden | XX | xx.x% | xx | xx.x% |
| | Amputation | XX | xx.x% | XX | xx.x% |
| SALVATION™ Midfoot Nail | Insulin Use | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ulcers | New | | Ulcer | |
| | | Ulcer | | Healing | |
| | Yes | XX | xx.x% | XX | xx.x% |
| | No | XX | xx.x% | XX | xx.x% |
| | Chronic Ulcer | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | New Deep Infection | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ankle Alignment | | | | |
| | Acceptable | | | XX | xx.x% |
| | Unacceptable | | | XX | xx.x% |
| | Not applicable | | | XX | xx.x% |
| | Current Status | | | | |
| | Walking | xx | xx.x% | XX | xx.x% |
| | Mobility with aids | XX | xx.x% | XX | xx.x% |




| Device | Factors | 1 Yea | r Visit | Final | Visit |
|---|---|---|---|---|---|
| | | N | % | N | % |
| | Wheelchair | XX | xx.x% | XX | xx.x% |
| | Bed ridden | XX | xx.x% | XX | xx.x% |
| | Amputation | XX | xx.x% | XX | xx.x% |
| SALVATION™ 3Di Plating | Insulin Use | | | | |
| System | | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ulcers | New | | Ulcer | |
| | | Ulcer | | Healing | |
| | Yes | XX | xx.x% | XX | xx.x% |
| | No | XX | xx.x% | XX | xx.x% |
| | Chronic Ulcer | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | New Deep Infection | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ankle Alignment | | | | |
| | Acceptable | | | XX | xx.x% |
| | Unacceptable | | | XX | xx.x% |
| | Not applicable | | | XX | xx.x% |
| | Current Status | | | | |
| | Walking | XX | xx.x% | XX | xx.x% |
| | Mobility with aids | XX | xx.x% | XX | xx.x% |
| | Wheelchair | XX | xx.x% | XX | xx.x% |
| | Bed ridden | XX | xx.x% | XX | xx.x% |
| | Amputation | XX | xx.x% | XX | xx.x% |
| <b>VALOR™ Nail</b> | Insulin Use | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ulcers | New | | Ulcer | |
| | | Ulcer | | Healing | |
| | Yes | XX | xx.x% | XX | xx.x% |
| | No | XX | xx.x% | XX | xx.x% |
| | Chronic Ulcer | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | New Deep Infection | | | | |
| | Yes | XX | xx.x% | | |
| | No | XX | xx.x% | | |
| | Ankle Alignment | | | | |
| | Acceptable | | | XX | xx.x% |
| | Unacceptable | | | XX | xx.x% |
| | Not applicable | | | XX | xx.x% |




| Device | Factors | 1 Yea | r Visit | Fina | al Visit |
|--------|-----------------------|-------|---------|------|----------|
| | | N | % | N | % |
| | <b>Current Status</b> | | | | |
| | Walking | XX | xx.x% | XX | xx.x% |
| | Mobility with aids | XX | xx.x% | XX | xx.x% |
| | Wheelchair | XX | xx.x% | XX | xx.x% |
| | Bed ridden | XX | xx.x% | XX | xx.x% |
| | Amputation | XX | xx.x% | XX | xx.x% |



**Table 3.4 Radiographic Assessment** 

| | | | Pre | Pre-onerative | ative | | | | H | Final Visit | sit | | | | Impr | Improvement | ent | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | п | mean | ps | min | max | 95% CI | u | mean | ps | mim | max | 95% CI | u | mean | ps | min | max | 95% CI |
| SALVATION™ 3Di Plating System | tem | | | | | | | - | | - | | | | | | | | |
| AP Meary's Angle | XX | x.xx | X.X | XX | XX | (xx.x, xx.x) | XX | xx.x | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Lateral Meary's Angle | XX | XXX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Talonavicular Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Cuboid height (mm) | XX | XXX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) |
| SALVATION™ External Fixation | on | | | | | | | | | | | | | | | | | |
| AP Meary's Angle | XX | XXXX | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Lateral Meary's Angle | XX | XXXX | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) |
| Talonavicular Meary's Angle | XX | XXXX | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) |
| Cuboid height (mm) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| SALVATION™ Fusion Bolts and Beams | ıd Be | ams | | | | | | | | | | | | | | | | |
| AP Meary's Angle | XX | XXXX | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) |
| Lateral Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Talonavicular Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | xx.x | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) |
| Cuboid height (mm) | XX | XXXX | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| SALVATIONT MIDFOOT NAIL | , | | | | | | | | | | | | | | | | | |
| AP Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Lateral Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Talonavicular Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Cuboid height (mm) | XX | XX.X | x.x | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Valor™ Nail | | | | | | | | | | | | | | | | | | |
| AP Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | X | XX.X | X.X | XX | XX | (xx.x, xx.x) | X | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Lateral Meary's Angle | XX | XX.X | X.X | XX | XX | (xx.x, xx.x) | X | XX.X | X.X | XX | XX | (xx.x, xx.x) | X | XX.X | X.X | XX | XX | (xx.x, xx.x) |
| Cuboid height (mm) | XX | XX.X | X.X | XX | X | (xx.x, xx.x) | X | XX.X | x.x | XX | XX | (xx.x, xx.x) | X | XX.X | X.X | X | XX | (xx.x, xx.x) |
| Talonavicular Meary's Angle | X | XX.X | X.X | XX | X | (XXX, XXX) | X | XX.X | X.X | XX | XX | (XXX, XXX) | X | XX.X | X.X | X | XX | (XX.X, XX.X) |

# stryker

# Statistical Analysis Plan for FINS (US20-SAL-001)

Table 4.1 Summary of All Adverse Events

| | SALVATION <sup>™</sup> Fusion Bolts ar Beams (N = xx) | ON™<br>Its and<br>Is | SALVATION™<br>MIDFOOT NAIL<br>(N = xx) | ION™<br>F NAIL<br>x) | SALVATION™<br>External Fixation<br>(N = xx) | ION™<br>ixation<br>x) | SALVATION™ 3Di<br>Plating System<br>(N = xx) | N™ 3Di<br>ystem | VALOR™ Nail<br>(N = xx) | "Nail<br>cx) |
|---|---|---|---|---|---|---|---|---|---|---|
| | Subjects | Event | Subjects | Event | Subjects | Event | Subjects | Event | Subjects | Event |
| Total | (%x.xx)xx | XX | xx(xx.x%) | XX | xx(xx.x%) | XX | (%x:xx)xx | XX | xx(xx.x%) | XX |
| Procedure-Related | (%x:xx)xx | XX | xx(xx.x%) | XX | (%x:xx)xx | xx | (%x:xx)xx | XX | (%x:xx)xx | xx |
| Device-Related | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | xx |
| Device Failure | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | xx |
| UADE | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX |
| Unanticipated AE | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX |
| Serious AE | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX |
| Hospitalization | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | xx(xx.x%) | xx |
| Death | (%x.xx)xx | xx | (%x.xx)xx | XX | (%x.xx)xx | xx | (%x:xx)xx | xx | xx(xx.x%) | xx |
| Required Treatment** | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX |
| Physical Therapy | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | xx |
| Medication | (%x:xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX |
| Surgery | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | xx |
| Other | (%x:xx)xx | XX | (%x.xx)xx | XX | (%x.xx)xx | XX | (%x:xx)xx | XX | (%x.xx)xx | xx |

# stryker

# Statistical Analysis Plan for FINS (US20-SAL-001)

Table 4.2 Device-related Adverse Events

| Surgery<br>date |
|------------------------------|
| UADE<br>(Y/N) |
| Device UADE<br>Failure (Y/N) |
| Event<br>Description |
| Onset<br>Days |
| ce(s) Device<br>Indication |
| Device(s) |
| Age Gender Devic |
| Age |
| Subject<br>ID |

Table 4.3 Serious Adverse Events

| Outcome |
|----------------------------------|
| SAE Onset Days Event Description |
| SAE Onset Days |
| Device<br>Indication |
| Device |
| Gender |
| Age |
| Subject ID |

**Certificate Of Completion** 

Envelope Id: 215FCFE3E56841B4B41B5DC7E89E9D7A

Subject: Complete with DocuSign: FINS US-20 SAL-001 Statistical Analysis Plan 6Jan2023-Final.pdf

Source Envelope:

Document Pages: 36

Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC-08:00) Pacific Time (US & Canada)

Status: Completed

Envelope Originator:

Jovi Quiton

jovelyn.quiton@stryker.com IP Address: 104.4.253.93

**Record Tracking** 

Status: Original

2/14/2023 5:36:56 AM

Holder: Jovi Quiton

jovelyn.quiton@stryker.com

Location: DocuSign

**Signer Events** 

David Fitch david.fitch@stryker.com

Security Level: Email, Account Authentication

(None)

**Signature** 

Signatures: 4

Initials: 0

DocuSigned by: David Fitch E1459B1F4E7B4D1..

Signature Adoption: Pre-selected Style

Using IP Address: 4.31.14.131

**Timestamp** 

Sent: 2/14/2023 5:41:29 AM Resent: 2/22/2023 7:16:09 AM Viewed: 2/22/2023 7:17:07 AM Signed: 2/22/2023 7:17:16 AM

**Electronic Record and Signature Disclosure:** 

Accepted: 9/20/2022 9:15:51 AM ID: 193d2803-eb49-4082-9f74-157c1f9d2a2e

Jovi Quiton

jovelyn.quiton@stryker.com Senior Manager, Statistics

Security Level: Email, Account Authentication

(None)

plyputon

DocuSigned by:

Monica Fleeman

9D851D9BB8FC415...

Signature Adoption: Uploaded Signature Image

Using IP Address: 104.4.253.93

Sent: 2/14/2023 5:41:30 AM Viewed: 2/22/2023 7:14:54 AM

Signed: 2/22/2023 7:15:03 AM

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

Monica Fleeman

monica.fleeman@stryker.com Sr. Clinical Study Manager

Stryker

Security Level: Email, Account Authentication

(None)

**Electronic Record and Signature Disclosure:** Accepted: 2/14/2023 6:23:25 AM

ID: 16e7aa87-dfcb-4baf-9f00-e3bcc981096f

Rebecca Gibson

Rebecca.Gibson@stryker.com Director, Clinical Operations

Stryker Corporation - Trauma & Extremitites Security Level: Email, Account Authentication

(None)

DocuSigned by: Kebecca Gibson B69B71B0C1FA437...

Signature Adoption: Pre-selected Style Using IP Address: 206.74.115.202

Signature Adoption: Pre-selected Style

Using IP Address: 76.214.178.82

Sent: 2/14/2023 5:41:29 AM Viewed: 2/14/2023 6:23:25 AM

Signed: 2/14/2023 6:23:31 AM

**Electronic Record and Signature Disclosure:** 

Accepted: 8/30/2022 7:58:43 AM

ID: ba2910e0-ad1a-4548-88ee-9a3a66121c1a

Sent: 2/14/2023 5:41:30 AM Viewed: 2/15/2023 4:25:45 PM Signed: 2/15/2023 4:28:44 PM

In Person Signer Events

Signature

**Timestamp** 

| Editor Delivery Events | Status | Timestamp |
|---|---|---|
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Notary Events Envelope Summary Events | Signature<br>Status | Timestamps |
| | - | · |
| Envelope Summary Events | Status | Timestamps |
| Envelope Summary Events Envelope Sent | Status Hashed/Encrypted | Timestamps 2/14/2023 5:41:30 AM |
| Envelope Summary Events Envelope Sent Certified Delivered | Status Hashed/Encrypted Security Checked | Timestamps 2/14/2023 5:41:30 AM 2/15/2023 4:25:45 PM |
| Envelope Summary Events Envelope Sent Certified Delivered Signing Complete | Status Hashed/Encrypted Security Checked Security Checked | Timestamps 2/14/2023 5:41:30 AM 2/15/2023 4:25:45 PM 2/15/2023 4:28:44 PM |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Jovi Quiton (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### How to contact Jovi Quiton:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: jovelyn.quiton@stryker.com

#### To advise Jovi Quiton of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at jovelyn.quiton@stryker.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Jovi Quiton

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to jovelyn.quiton@stryker.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Jovi Quiton

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to jovelyn.quiton@stryker.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Jovi Quiton as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Jovi Quiton during the course of your relationship with Jovi Quiton.